CLINICAL TRIAL: NCT02758587
Title: A Phase I/IIA Study to Assess Safety, Tolerability and Preliminary Activity of the Combination of FAK (Defactinib) and PD-1 (Pembrolizumab) Inhibition in Patients With Advanced Solid Malignancies (FAK-PD1)
Brief Title: Study of FAK (Defactinib) and PD-1 (Pembrolizumab) Inhibition in Advanced Solid Malignancies (FAK-PD1)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Cancer Research UK (Other); Merck Sharp & Dohme LLC (Industry); Verastem, Inc. (Industry); University of Edinburgh (Other); University of Southampton (Other); University of Leicester (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN15ON133; 2015-003928-31 (EudraCT Number)
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-small-cell Lung; Mesothelioma; Pancreatic Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma; Pancreatic Neoplasms | interventions — defactinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose - escalation (Experimental): Does-escalation in an "all-comers" phase I population, with treatment-refractory advanced solid malignancies, unselected by tumour type. Two cohorts of up to evaluable 6 patients in each:
  * Cohort 1: 200mg (IV) pembrolizumab every 3 weeks; plus 200mg (oral) defactinib twice daily
  * Cohort 2: 200mg (IV) pembrolizumab every 3 weeks; plus 400mg (oral) defactinib twice daily
  Interventions:
  * Drug: Defactinib
  * Drug: Pembrolizumab
  Interventions: Drug: Defactinib; Drug: Pembrolizumab
- Pancreatic (Experimental): Pancreatic expansion for response assessment (single arm). Optional paired biopsies prior to treatment and after 14 days of treatment. All would have concurrent therapy with pembrolizumab + defactinib (VS-6063) from the start (c.f. NSCLC & mesothelioma expansions below). 15 evaluable patients with an interim futility assessment for clinical response and tolerability when data available from 6
  Interventions: Drug: Defactinib; Drug: Pembrolizumab
- NSCLC (Experimental): NSCLC paired-biopsy expansion for tissue biomarkers. Mandatory biopsies prior to treatment and after around 14 days of treatment. 1:1 randomised split of patients having their mandatory on-treatment biopsy after concurrent therapy, or after a defactinib (VS-6063) monotherapy run-in. 16 evaluable patients with an interim futility assessment for clinical response and tolerability when data available from 11.
  Interventions: Drug: Defactinib; Drug: Pembrolizumab
- Mesothelioma (Experimental): Mesothelioma paired-biopsy expansion for tissue biomarkers. Mandatory biopsies prior to treatment and around 14 days of treatment. 1:1 randomised split of patients having thier on-treatment biopsy after concurrent therapy, or after defactinib (VS-6063) monotherapy run-in. 16 evaluable patients with an interim futility assessment for clinical response and tolerability when data available from 11.
  Interventions: Drug: Defactinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Defactinib — cross reference with arm/group descriptions
  Other Names: VS-6063
Drug: Pembrolizumab — cross reference with arm/group descriptions
  Other Names: Keytruda and MK-3475

SUMMARY:
This study will explore whether defactinib (a FAK inhibitor) can be safely and tolerably combined with pembrolizumab (a PD-1 inhibitor) and will look for early indications of improved anticancer immunotherapy. It will focus on three key cancers, all in clear need of improved therapies - NSCLC, pancreatic cancer and mesothelioma.

DETAILED DESCRIPTION:
Programmed cell death receptor 1 (PD-1) blockade is a well-tolerated novel cancer immunotherapy with monotherapy response rates of 20-50% in tumour types such as bladder, melanoma, renal and non-small cell lung cancer (NSCLC), along with durable benefit. However, other tumour types (such as pancreatic cancer) have been poorly responsive and it is likely that the activity of PD-1 blockade is limited in many patients by the presence of additional immunosuppressive tumour microenvironment interactions. The investigators have recently shown in preclinical studies that Focal Adhesion Kinase (FAK) inhibition can re-model multiple aspects of the tumour immune microenvironment, shifting the balance from inhibitory Tregs, TAMs, CAFs & MDSCs, to one which supports an active CD8+ T cell adaptive immune response, suitable for synergistic anti-PD-1 therapy.

The current clinical study will explore whether FAK inhibition (defactinib/VS-6063) can be safely and tolerably combined with PD-1 blockade (pembrolizumab), with early indications of improved anticancer immunotherapy from this novel combination. The investigators will focus on three key tumour types, all cancers in clear need of improved therapies. NSCLC, aiming to augment the moderate monotherapy activity of PD-1 blockade; pancreatic cancer, aiming to release immunological activity in this otherwise resistant cancer; and, finally, mesothelioma, where emerging data suggests both agents may have monotherapy activity, including a potential additional mode of action via synthetic lethality of FAK inhibition in the ~50% of mesothelioma with NF2 mutation.

Phase I/IIa clinical study of defactinib (VS-6063, FAK inhibitor) in combination with pembrolizumab (anti-PD-1) therapy, initially in an "all-comers" dose escalation phase, and subsequently in expansion cohorts at the optimal doses in patients with: (a) pancreatic cancer; (b) NSCLC; and (c) mesothelioma. Safety, tolerability and clinical activity will be explored, as well as extensive translational work to characterise the biological effects and explore potential predictive and pharmacodynamic biomarkers.

PHASE I

Dose-escalation in an "all-comers" phase I population, with treatment-refractory advanced solid malignancies, unselected by tumour type as follows:

Cohorts 200 mg (IV) pembrolizumab every 3 weeks: plus 200 mg (oral) defactinib twice daily 200 mg (IV)pembrolizumab every 3 weeks: plus 400 mg (oral) defactinib twice daily

PHASE II

Expansions in pancreatic ductal adenocarcinoma, non-small cell lung cancer & mesothelioma (each 15-16 evaluable patients).

Pancreatic

Pancreatic expansion for response assessment (single arm). Optional paired biopsies prior to treatment and after 14 days of treatment. Concurrent therapy with pembrolizumab + defactinib (VS-6063) from the start (c.f. NSCLC & mesothelioma expansions below). 15 evaluable patients with an interim futility assessment for clinical response and tolerability when data available from 6.

* Classic "stromal" cancer, where the tumour microenvironment is believed to limit the activity of multiple agents. However broad preclinical data for various approaches to re-modelling the tumour microenvironment to permit immunotherapy.
* Minimal single-agent anti-PD-1/PD-L1 activity, explores hypothesis of conversion to sensitivity and predictive biomarkers for this.

NSCLC

NSCLC paired-biopsy expansion for tissue biomarkers. Mandatory biopsies prior to treatment and after around 14 days of treatment. 1:1 randomised split of patients having their on-treatment biopsy after concurrent therapy, or after a defactinib (VS-6063) monotherapy run-in. 16 evaluable patients with an interim futility assessment for clinical response and tolerability when data available from 11.

* Moderate single-agent anti-PD-1/PD-L1 activity explores hypothesis of amplification of sensitivity and predictive biomarkers for this.
* Paired-biopsy assessment of proof of mechanism biomarkers (FAK signalling, tumour immune microenvironment).

Mesothelioma

Mesothelioma paired-biopsy expansion for tissue biomarkers. Mandatory biopsies prior to treatment and after around 14 days of treatment. 1:1 randomised split of patients having their on-treatment biopsy after concurrent therapy, or after a defactinib (VS-6063) monotherapy run-in). 16 evaluable patients with an interim futility assessment for clinical response and tolerability when data available from 11.

* Emerging single-agent immune checkpoint, as well as potential FAK-inhibitor activity, explores hypothesis of multi-modal combination activity (microenvironment, checkpoint and synthetic lethality), as well as predictive biomarkers for this.
* Paired-biopsy assessment of proof of mechanism biomarkers (FAK signalling, tumour immune microenvironment).

ELIGIBILITY:
Inclusion Criteria:

All Patients:

* Informed, written consent
* Male or female, aged 18 years or older at the time consent is given
* ECOG performance status 0 or 1, with no deterioration over the previous 2 weeks
* Life expectancy of at least 3 months
* Measurable disease according to irRECIST criteria, with at least one measurable lesion that has objectively progressed since (or on) any previous therapy
* Adequate bone marrow, liver and renal function on blood investigations within 7 days prior to treatment initiation
* Patients must have been offered all appropriate standard-of-care treatments (or all those indicated before anti-PD-1/PD-L1 therapy, if licensed)
* Patients must agree to use adequate contraceptive measures for the course of the study through 120 days after the last dose of study medication
* Women of child-bearing potential must have a negative pregnancy test within 72 hours prior to start of dosing
* Consent to supply any available archival tissue

Dose escalation (Phase I):

* Pathological diagnosis of any advanced solid tumour type, with confirmation that a tissue sample (core biopsy or resected specimen) is available

Pancreatic expansion (Phase IIa):

* Pathological diagnosis of pancreatic ductal adenocarcinoma with confirmation that a tissue sample (core biopsy or resected specimen) is available

NSCLC expansion (Phase IIa):

* Pathological diagnosis of non-small cell lung cancer (NSCLC)
* Lesion suitable for repeat biopsy
* Baseline biopsy containing tumour material during eligibility
* Consent for paired biopsies on study

Mesothelioma expansion (Phase IIa):

* Pathological diagnosis of mesothelioma
* Lesion suitable for repeat biopsy
* Baseline biopsy containing tumour material during eligibility
* Consent for paired biopsies on study

Exclusion Criteria:

All patients:

* An additional invasive cancer in the last 5 years (other than treated and controlled localised non-melanoma skin cancer or cervical carcinoma-in-situ, or indolent prostate cancer that has been stable for > 1 year)
* Any central nervous system metastases unless treated and asymptomatic, as well as stable on imaging and not requiring steroids in the preceding 4 weeks
* Any interventional studies, systemic cancer therapies or monoclonal antibodies in the preceding 4 weeks (6 weeks for mitomycin C and nitrosureas)
* Any live vaccines in the preceding 4 weeks
* Systemic immunosuppressive agents in the preceding 2 weeks. Immunosuppressive agents include steroids such as prednisolone (doses ≥ 15 mg daily) or dexamethasone (doses ≥ 2 mg daily).

Replacement therapy (e.g. physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency etc) is not considered a form of systemic treatment

* Diagnosis of immunodeficiency
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known interstitial lung disease or active, non-infectious pneumonitis
* Known history of Tuberculosis (TB), Human Immunodeficiency Virus (HIV) or active Hepatitis B or C
* Other severe or uncontrolled systemic diseases (e.g. uncontrolled hypertension, recent myocardial infarction, organ failure or active infection)
* Residual (non-laboratory) toxicities greater than grade 1 (CTCAE v4.03) from previous therapies despite optimal supportive therapy, including fatigue, anorexia, nausea or diarrhoea, but with the exception of alopecia
* Pregnancy or lactation
* Limited ability to swallow or absorb oral medications
* Hypersensitivity to defactinib (VS-6063), pembrolizumab or excipients (including L-histidine, L-histidine hydrochloride monohydrate, sucrose or polysorbate 80)
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Previous treatment with an anti-PD-1 or anti-PDL1 agent
* Previous severe or life-threatening skin adverse reaction with other immune-stimulatory anticancer agents
* Current solid organ transplant recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) using CTCAE v4.03 (to determine dose limiting toxicities (DLTs) and maximum tolerated dose (MTD)) | 6 months
  Evaluate the tolerability profile and optimal dose of defactinib in combination with pembrolizumab, using CTCAE v4.03 Adverse Event recording.

SECONDARY OUTCOMES:
Objective response rate (ORR), using best objective response by irRECIST | 3 years
  Evaluate the response rate, by irRECIST, of the combination of defactinib and pembrolizumab in patients with advanced solid malignancies.
Duration of response (DoR) | 3 years
  Evaluate the duration of responses, by irRECIST, of the combination of defactinib and pembrolizumab in patients with advanced solid malignancies. Duration will be measured from the first scan showing radiological response (CR or PR), until (irRECIST confirmed) progression.
Progression free survival (PFS) | 3 years
  Evaluate progression free survival of the combination of defactinib and pembrolizumab in patients with advanced solid malignancies. Duration will be measured from enrolment, until (irRECIST confirmed) progression.
Change in FAK Y397 phosphorylation | 2 weeks
  change in FAK Y397 phosphorylation between baseline biopsy and a repeat biopsy afer 2 weeks of therapy
Change in immune cell infiltrate | 2 weeks
  change in immune cell infiltrate between baseline biopsy and a repeat biopsy after 2 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Symeonides, Principal Investigator — Edinburgh Cancer Research Centre, University of Edinburgh, Western General Hospital, Edinburgh EH4 2XR; Jeff Evans, Principal Investigator — Beatson West of Scotland Cancer Centre, 1053 Great Western Road, Glasgow G12 0YN; Christian Ottensmeier, Principal Investigator — Cancer Research UK Centre, Southampton University Hospitals and University of Southampton, Southampton SO16 6YD; Dean Fennell, Principal Investigator — Department of Cancer Studies, University of Leicester, Leicester Royal Infirmary, Leicester LE2 7LX; Vicky Coyle, Principal Investigator — Belfast Health and Social Care Trust, Cancer Centre, Lisburn Road, Belfast BT9 7BL
Locations (5):
- United Kingdom (5):
  - Belfast Health and Social Care Trust, Cancer Centre, Lisburn Road, Belfast
  - Edinburgh Cancer Research Centre, Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Department of Cancer Studies, University of Leicester, Leicester Royal Infirmary, Leicester
  - Cancer Research UK Centre, Southampton University Hospitals and University of Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fard D, Giraudo E, Tamagnone L. Mind the (guidance) signals! Translational relevance of semaphorins, plexins, and neuropilins in pancreatic cancer. Trends Mol Med. 2023 Oct;29(10):817-829. doi: 10.1016/j.molmed.2023.07.009. Epub 2023 Aug 17. PMID 37598000